CLINICAL TRIAL: NCT07086755
Title: Vadadustat for the Treatment of Nonintubated Acute Respiratory Distress Syndrome Due to Pathogen-Associated Lung Injury
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bentley J. Bobrow (Other)
Collaborators: Akebia Therapeutics Inc. (Unknown)
Responsible Party: Sponsor-Investigator, Bentley J. Bobrow, Professor, The University of Texas Health Science Center, Houston
Organization: The University of Texas Health Science Center, Houston (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC-MS-22-0260
Record Dates: First submitted 2025-07-18; First posted 2025-07-25 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Nonintubated Acute Respiratory Distress Syndrome (ARDS); Pathogen-associated Lung Injury
MeSH Terms: interventions — vadadustat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Vadadustat 900mg (Experimental)
  Interventions: Drug: Vadadustat 900mg
- Vadadustat 1200mg (Experimental)
  Interventions: Drug: Vadadustat 1200mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vadadustat 900mg — Participants will receive 900mg vadadustat (as oral tablets) for 14 days or until the date of discharge, whichever comes first, at approximately the same time each day without regard for timing of meals.
  Arms: Vadadustat 900mg
Drug: Vadadustat 1200mg — Participants will receive 1200mg vadadustat (as oral tablets) for 14 days or until the date of discharge, whichever comes first, at approximately the same time each day without regard for timing of meals.
  Arms: Vadadustat 1200mg
Drug: Placebo — Participants will matching placebo (as oral tablets) for 14 days or until the date of discharge, whichever comes first, at approximately the same time each day without regard for timing of meals.
  Arms: Placebo

SUMMARY:
The objective of this study is to assess the efficacy and safety of vadadustat for treating hospitalized patients with nonintubated Acute Respiratory Distress Syndrome (ARDS) secondary to pathogen-associated lung injury.

ELIGIBILITY:
Inclusion Criteria:

-Meets the definition of nonintubated ARDS per the 2024 Global Definition of ARDS that includes all the following (2A-2D):

* 2A. Risk factors and origin of pulmonary edema: Precipitated by an acute predisposing risk factor, specifically from a suspected pathogen-associated etiology such as pneumonia* or non-pulmonary infection** [*Pneumonia defined as known or suspected based on treating physician documentation or discussion, OR both of the following criteria: 1) Chest radiography with new infiltrates, consolidation, or cavitation and (2) Clinical signs of pneumonia (new cough, sputum, fever, or white blood cells (WBC) > 12,000)] [**Non-pulmonary infection defined as suspected or proven infection meeting any of the following criteria: treating clinician suspects a viral, bacterial, or fungal infection, or cultures ordered in the past 24h or positive cultures within 1 week; or orders for antimicrobial medication.]
* 2B. Oxygenation: PaO2:FIO2 ≤ 300 mm Hg or SpO2:FIO2 ≤ 315 (if SpO2 ≤ 97%) on High-Flow Nasal Oxygen (HFNO) with flow of ≥ 30 L/min or non-invasive ventilation (NIV)/continuous positive airway pressure (CPAP) with at least 5 cm H2O end-expiratory pressure
* 2C. Timing: Acute onset or worsening of hypoxemic respiratory failure within 1 week of the estimated onset of the predisposing risk factor or new or worsening respiratory symptoms.
* 2D. Chest imaging: Chest infiltrates on radiography and computed tomography or B lines and/or consolidations on ultrasound not fully explained by effusions, atelectasis, or nodules/masses.

Exclusion Criteria:

* Hypersensitivity to vadadustat or any of its excipients
* Placed on mechanical ventilation before randomization
* Patients on home oxygen therapy
* Time since hospital admission order placed >72 hours
* Hemoglobin above the gender-specific upper limit of normal (ULN) at randomization: 16 grams/deciliter (g/dL) for females and 18 g/dL for males
* Patients with Aspartate transferase (AST) or Alanine aminotransferase (ALT) levels >5 times the upper limit of normal
* Patients with AST or ALT levels >3 times the upper limit of normal along with a total bilirubin elevation of >2 times the upper limit of normal.
* Patients who have erythrocytosis or polycythemia vera
* Patients with uncontrolled hypertension
* Patients with active malignancy
* Patients with liver cirrhosis or active, acute liver disease
* Patients taking erythropoiesis-stimulating agents
* Patient taking probenecid, rifampicin, gemfibrozil, or teriflunomide
* Women who are pregnant or breastfeeding, or positive pregnancy test before randomization
* Patients who are prisoners
* Patients who are currently enrolled in any other interventional clinical trial
* Patients who have any prior history of arterial or venous thromboembolism within the past 3 months
* Patients with a history of myocardial infarction, cerebrovascular event, or acute coronary syndrome within the past 3 months
* Patients with known or suspected tuberculosis infection
* Moribund patient not expected to survive 48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2025-10-23 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Win ratio for hierarchical composite endpoint based on death, duration of mechanical ventilation or ECMO, and duration of high-flow nasal oxygenation or non-invasive ventilation | from the time of enrollment to 28 days after enrollment
  The primary outcome is a hierarchical composite endpoint with 3 components: Death (yes or no); Duration of mechanical ventilation (MV) or extracorporeal membrane oxygenation (ECMO) in days; and Duration of high-flow nasal oxygenation (HFNO) or noninvasive ventilation (NIV) in days. Data will be reported as a Win Ratio, which quantifies the relative benefit of treatment compared to control. The Win Ratio is calculated from all pairwise comparisons of each patient in the treatment group compared with each patient in the control group, using the following formula: Win Ratio = Number of Wins/Number of Losses. Number of Wins is defined as: The count of pairs where the treatment group patient has a better outcome than the control group patient. Number of Losses is defined as: The count of pairs where the control group patient has a better outcome than the treatment group patient.

SECONDARY OUTCOMES:
Number of deaths | from the time of enrollment to 28 days after enrollment
Duration of mechanical ventilation (MV) or extracorporeal membrane oxygenation (ECMO) in days | from the time of enrollment to 28 days after enrollment
Duration of high-flow nasal oxygenation (HFNO) or noninvasive ventilation (NIV) in days | from the time of enrollment to 28 days after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Paul Potnuru, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No